CLINICAL TRIAL: NCT05103696
Title: Safety and Efficacy of Remazolam in Gastroenteroscopy in Elderly Patients
Brief Title: A Comparative Study of Rimazolam and Propofol Combined With Etomidate in Gastroenteroscopy in Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Yi Feng, MD, Chief of Anesthesiology department, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2021PHB002-001
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Elderly Patients; Gastrointestinal Endoscopy; Remimazolam Besylate; Etomidate Combined With Propofol
Keywords: Remimazolam Besylate; Etomidate combined with propofol; Gastrointestinal Endoscopy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): Patients received remimazolam to maintain sufficient sedation (sufficient sedation as judged by MOAA/S ≤ 4 for 3 consecutive measurements) during endoscopy procedure. And patients were injected remifentanil 0.3μg/kg (infusion time > 1min) at the first time，When the analgesia was insufficient, Remifentanil can be added according to the situation.
  Interventions: Drug: Remimazolam Besylate
- EP group (Active Comparator): Patients received Etomidate combined with propofol to maintain sufficient sedation (sufficient sedation as judged by MOAA/S ≤ 4 for 3 consecutive measurements) during endoscopy procedure. And patients were injected remifentanil 0.3μg/kg (infusion time > 1min) at the first time.When the analgesia was insufficient,Remifentanil can be added according to the situation
  Interventions: Drug: etomidate combined with propofol

INTERVENTIONS:
Drug: Remimazolam Besylate — Remazolam 7mg for the first time (push time 1min), 2.5mg can be added after 2min according to MOAA/S score, no more than 5 times within 15min
  Arms: Remimazolam group
Drug: etomidate combined with propofol — Etomidate 0.1mg/kg+1% propofol 0.5mg/kg for the first time ,etomidate0.05mg/kg+ 1% propofol 0.25 mg/kg can be added according to MOAA/S score
  Arms: EP group

SUMMARY:
Studies have shown that etomidate combined with propofol in gastroscopy has high safety and lower incidence of hypoxia and hypotension, suggesting the advantages of etomidate combined with propofol in elderly patients.

Remimazolam Besylate is a 1.1 class new drug that acts on GABA receptors and is metabolized by plasma esterase with fast metabolism time, only 1/7 of midazolam, which may be more suitable for elderly patients. Therefore, this study intends to explore the safety and effectiveness of two sedation schemes in gastroenteroscopy for elderly patients.

DETAILED DESCRIPTION:
Before starting the endoscopy procedures, patients were randomly assigned to either Remimazolam Besylate group or propofol combined with etomidate group. The onset time, recovery time, vital signs, postoperative recovery, cognitive function and adverse events were compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with asAI-II indications for painless gastroenteroscopy and receiving diagnostic or therapeutic gastroenteroscopy;
2. Aged 60-75, body mass index (BMI) 19-28 kg/m2, Systolic blood pressure of 90-140mmHg, diastolic blood pressure of 50-90mmHg, resting heart rate of 50-100bpm and blood pulse oxygen saturation ≥95%

Exclusion Criteria:

1. Those who are refused to be included;
2. Those who are allergic to the drugs used in this study;
3. Epilepsy and other mental illnesses, a history of addiction such as opiates and other analgesics and/or tranquilizers (hypnotics);
4. Severe lung infection or upper respiratory tract infection;

7. Sleep apnea syndrome, difficult airway (Mallampati score of 3 or 4) or asthma status; 8. Advanced cancer accompanied by extensive intra-abdominal metastasis;

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
induction time | day 0
  The time from the beginning of the drug injection to the time when the patient does not respond to the verbal call
Recovery time | day 0
  First of 3 consecutive MOAA/S scores of 5 after the last injection of study drug
Modified Observer's Assessment of Alertness/Sedation[MOAA/S] | day 0
  MOAA/S score ranges from 0 to 5 points, 0 point means patients do not respond to noxious stimulation; 5 point means patients responds readily to name spoken in normal tone. When the Modified Observer's Assessment of Alertness/ Sedation [MOAA/S] ≤4 that patients are sufficiently sedated.
Observation time in the PACU | day 0
  the time interval between "endoscope removal" and "departure from the recovery room" （PADS score≥9）

SECONDARY OUTCOMES:
Simple Intelligence Assessment Scale (mini-cog) | Every 4 hours, up to 1 week
  1. Ask the subjects to listen carefully and memorize 3 unrelated words, and then repeat (Apple, Watch, Coin);
  2. Ask the subjects to draw the shape of the clock on a blank sheet of paper, and give the subject a time to mark it on the clock (the CDT of the clock drawing test is correct; it can correctly indicate the sequence of the digits and display the given Fixed time);
  3. Ask the subject to say the 3 words given previously.
Drug dosages | day 0
  The total single dosage of remimazolam , propofol, etomidate，remifentanil and tosilate.
Patient overall satisfaction and surgeon satisfaction score | day 0
  The patient's overall satisfaction score and surgeon satisfaction score were evaluated by 1-10 points (1mm=completely dissatisfied, 100mm=completely satisfied).
Visual analogue scale (VAS) | day 0
  The visual analogue scale (VAS) score ranges from 0 to 10 points (0mm means patients feel no pain, 100mm means patients feel the most severe pain imaginable)
Level of hypoxia | day 0
  Oxygen saturation <90% for more than 1 minute #that share a common Unit of Measure in（%）
Respiratory depression | day 0
  Respiratory rate < 8 breaths per minute ,that share a common Unit of Measure in（times）
Rate of nause、vomiting、 dizziness、hiccups、 cough choking 、body movement | Within 24 hours
  Rate of nause、vomiting、 dizziness、hiccups、 cough choking 、body movement in （%） Rate of coughing and vomiting in（%）
Supine heart rate[HR] | day 0
  Supine heart rate[HR] in (times)
Systolic, diastolic, blood pressure | day 0
  Systolic, diastolic, blood pressure in(mmHg)
Assessment of pulse oximetry measurements[SpO2] | day 0
  Assessment of pulse oximetry measurements[SpO2]in(%)
Respiration rate[RR] | day 0
  Respiration rate[RR] in (times)
End-tidal carbon dioxide [EtCO2] | day 0
  End-tidal carbon dioxide [EtCO2] in (%）

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No